CLINICAL TRIAL: NCT06093399
Title: Stimulation of the Thalamus to Ameliorate Parkinsonian Speech Disfluencies: Pilot Study
Brief Title: Parkinsonian Sutter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Professor of Neurosurgery, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H23-02962
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Parkinson's Disease Stutter
Keywords: Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will act as their own control. Each individual's stutter will be assessed with DBS system OFF (control) and DBS ON (treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Simulation (DBS) System (Experimental): The DBS device will be turned on to compare stutter to when the device was off (which would be the control).
  Interventions: Device: System ON; Device: System OFF

INTERVENTIONS:
Device: System ON — The DBS system will be turned on, and the individual's stutter will be assessed.
Device: System OFF — The DBS system will be turned off, and the individual's stutter will be assessed.

SUMMARY:
The research team aims to provide evidence of Parkinsonian (PD) Stutter management by addressing the primary neurological issue in this disorder using Deep Brain Stimulation (DBS). The team proposes to perform unilateral DBS on 3 patients with PD stutter refractory to intensive speech therapy, to determine a response in their PD stutter. The assessments will be double-blinded. The investigators will use the outcome of this case series to determine the feasibility and details of a larger randomized controlled trial.

DETAILED DESCRIPTION:
Purpose: The purpose is to assess if dominant thalamic Deep Brain Stimulation (DBS) is an effective treatment for Parkinsonian stutter. Functional magnetic resonance imaging (MRI) will detect brain dominance before surgery. The research team will assess whether dominant thalamic DBS is preferable for stutter treatment.

Hypothesis: The research team hypothesizes that dominant thalamic neuromodulation with DBS effectively treats PD stutter.

Justification:

The investigators initially began investigating the possibility of treatment of Stutter with DBS when they had a patient whose stutter serendipitously improved following thalamic DBS for tremor. The patient had severe tremor requiring bilateral thalamic DBS; he coincidentally had stutter. Post-operatively, the patient noted that he had had marked improvement in his tremor as well as his stutter. This prompted a literature search, where the investigators found that this has previously been reported in one other patient. Previous investigations of spasmodic dysphonia show that speech (similar to language) is lateralized in most patients, and that unilateral treatment of the dominant hemisphere is as beneficial as bilateral treatment.

Objectives: The objective is to perform a case series of three patients to assess feasibility and determine design of a future, larger study. If there is an appreciable reduction in stuttering with dominant stimulation, a larger unilateral (dominant) thalamic study can be undertaken. The magnitude of effect determined by this pilot trial will allow for a power calculation for the future study.

Research Design:

Pre-operatively, patients will complete "The One Page Stuttering Assessment," Overall Assessment of the Speaker's Experience of Stuttering (OASES), Voice-related Quality of Life (VRQoL), Beck Depression Inventory version II (BDI-II), and Montreal Cognitive Assessment (MoCA). Patients will then have a functional MRI scan and unilateral thalamic DBS systems implanted. The patient will be randomized to either the DBS on or DBS off group and complete the "One Page Stutter Assessment," OASES and VRQoL on both settings. After 6 months, an unblinded phase follows until the end of the study 12 months after surgery. At the end of the 12 month post-op, participants will complete the OASES, VRQoL, "One Page Stutter Assessment," MoCA and BDI-II.

Statistical Analysis: The primary outcome will be PD stutter severity, as assessed by the One-Page Sutter Assessment. Outcomes will be statistically compared by a Wilcoxon analysis for paired nonparametric measures with a significance set at P<0.05. Secondary outcomes will be the quality of life measures, Voice Related Quality of Life (VRQoL) and Overall Assessment of the Speaker's Experience of Stuttering (OASES), as well as the Montreal Cognitive Assessment (MoCA), and Beck Depression Inventory version II (BDI-II).

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 19 and 80 years old
* Individuals with persistent PD stutter

Exclusion Criteria:

* Patients with mild symptoms.
* Patients who have a neurodegenerative disease.
* Patients with a bleeding diathesis.
* non English speaking patients

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of One-Page Suttering Assessment from Baseline to Post-Operation | One-Page Stutter Assessment will be reported by the patients preoperatively, after three months of blinded DBS-ON and DBS-OFF, and then again after 6 months unblinded DBS-ON
  Objectively assesses individual's stutter. Divide the number of instances of stuttering by the number of syllables in the sample and multiply by 100 to obtain the percentage of stuttered syllables.

SECONDARY OUTCOMES:
Change of Voice Related Quality of Life (VRQoL) from Baseline to Post-Operation | V-RQOL will be reported by the patients preoperatively, after three months of blinded DBS-ON and DBS-OFF, and then again after 6 months unblinded DBS-ON
  A 10-question, 5 point rating scale assessment, with higher scores reflecting a worse subjective voice-related quality of life.
Change of Overall Assessment of the Speaker's Experience of Stuttering (OASES) from Baseline to Post-Operation | OASES will be reported by the patients preoperatively, after three months of blinded DBS-ON and DBS-OFF, and then again after 6 months unblinded DBS-ON
  5-point scale that indicates the amount of adverse impact a person experiences due to stuttering, with higher scores indicating higher levels of negative impact.